CLINICAL TRIAL: NCT06346067
Title: A Randomized, Open-label Phase III Study in Patients With Previously Treated Unresectable or Metastatic NRAS Mutant Cutaneous Melanoma Comparing the Combination of Naporafenib + Trametinib to Physician's Choice of Therapy (Dacarbazine, Temozolomide or Trametinib Monotherapy) With a Dose Optimization lead-in [SEACRAFT-2]
Brief Title: A Study to Assess Naporafenib (ERAS-254) Administered With Trametinib in Patients With NRAS-mutant Melanoma (SEACRAFT-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-254-02
Record Dates: First submitted 2024-03-17; First posted 2024-04-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Advanced or Metastatic NRAS-mutant Melanoma
Keywords: Melanoma; NRAS Mutant; Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — naporafenib; Dacarbazine; Temozolomide; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1 Dose selection Lead-in Arm 1 (Experimental): Naporafenib + Trametinib Naporafenib (ERAS-254) 100 mg administered orally twice daily (BID) Trametinib 1 mg once daily (QD)
  Interventions: Drug: Naporafenib; Drug: Trametinib
- Stage 1 Dose selection Lead-in Arm 2 (Experimental): Naporafenib + Trametinib Naporafenib (ERAS-254) 400 mg administered orally twice daily (BID) Trametinib 0.5 mg once daily (QD)
  Interventions: Drug: Naporafenib; Drug: Trametinib
- Stage 1 Dose selection Lead-in Arm 3 Trametinib monotherapy (Active Comparator): Trametinib 2 mg once daily (QD)
  Interventions: Drug: Trametinib
- Stage 2 Arm A (Experimental): Naporafenib + Trametinib Naporafenib (ERAS-254) BID oral administration with Trametinib QD at the dose selected in Stage 1
  Interventions: Drug: Naporafenib; Drug: Trametinib
- Stage 2 Arm B - Physician's Choice (Active Comparator): * Dacarbazine 1000 mg/m2 intravenously (IV) on Day 1 of each 21-day cycle OR
  * Temozolomide 200 mg/m2/day PO on Day 1 to Day 5 of each 28-day cycle OR
  * Trametinib monotherapy, 2 mg PO QD
  Interventions: Drug: Dacarbazine; Drug: Temozolomide; Drug: Trametinib

INTERVENTIONS:
Drug: Naporafenib — Naporafenib (ERAS-254) is an experimental Pan-Raf inhibitor
  Other Names: ERAS-254; LXH254
  Arms: Stage 1 Dose selection Lead-in Arm 1; Stage 1 Dose selection Lead-in Arm 2; Stage 2 Arm A
Drug: Dacarbazine — Dacarbazine IV - Day 1
  Other Names: DTIC
  Arms: Stage 2 Arm B - Physician's Choice
Drug: Temozolomide — Temozolomide 200 mg/m2/day PO on Day 1 to Day 5 of each 28-day cycle
  Other Names: Temodar; TMZ
  Arms: Stage 2 Arm B - Physician's Choice
Drug: Trametinib — Trametinib is an FDA approved anticancer medication that targets MEK1 and MEK2.
  Other Names: Mekinist

SUMMARY:
Stage 1: To select the optimal dose of naporafenib + trametinib to be studied in Stage 2.

Stage 2: To compare progression free survival (PFS) and overall survival (OS) for patients with NRAS-mutant (NRASm) melanoma who are randomized to receive the combination of naporafenib + trametinib to that of patients who are randomized to physician's choice of therapy (dacarbazine, temozolomide, or trametinib monotherapy).

DETAILED DESCRIPTION:
SEACRAFT-2 is a global, Phase III, open-label, randomized study to assess the efficacy and safety of naporafenib administered with trametinib compared to physician's choice of therapy (dacarbazine, temozolomide, or trametinib monotherapy) in patients with unresectable or metastatic NRAS mutant melanoma who have progressed on, or are intolerant to, an anti-programmed death-1 ligand 1 (PD 1/L1)-based regimen. The study will consist of 2 stages: dose optimization in Stage 1 and the Phase 3 portion in Stage 2.

A total of approximately 470 eligible patients will be randomized to receive study drug(s) in this study across 2 stages.

ELIGIBILITY:
Key Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age ≥ 18 years
3. Histologically or cytologically confirmed unresectable or metastatic cutaneous (includes acral) melanoma.
4. Documentation of an NRAS mutation (tumor tissue or blood) prior to first dose of study drug(s) as determined locally with an analytically validated assay in a certified testing laboratory.
5. Archival tumor tissue collected within 5 years prior to enrollment must be confirmed to be available at the time of Screening, which may be submitted before or after enrollment for exploratory biomarker analysis.
6. Must have received an anti-PD-1/L1 based regimen (monotherapy or combination). Patient must have documented disease progression either while receiving therapy or within 12 weeks of last dose of the most recent anti-PD-1/L1 based regimen; the patient is eligible if they have received other therapies between the most recent anti-PD-1/L1 based regimen and enrollment.
7. ECOG performance status 0, 1 or 2
8. Presence of at least 1 measurable lesion according to RECIST v1.1
9. Able to swallow oral medication.

Key Exclusion Criteria:

1. Patients with uveal or mucosal melanoma
2. Prior therapy with an ERK-, MEK-, RAF-, or RAS-inhibitor
3. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug(s) (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
4. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndrome)
5. LVEF <50%
6. Symptomatic CNS metastases that are neurologically unstable. Patients with controlled CNS metastases are eligible.
7. Patients receiving treatment with herbal medicine known to cause liver toxicity, which cannot be discontinued 7 days prior to first dose of study drug(s) and for the duration of the study.
8. Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Stage 1:To select the optimal dose of naporafenib + trametinib to be studied in Stage 2 | Assessed up to 6 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs
Stage 1:To select the optimal dose of naporafenib + trametinib to be studied in Stage 2 | Assessed up to 6 months from time of first dose
  Objective response rate (ORR) based on assessment of radiographic imaging RECIST v1.1
Stage 1:To select the optimal dose of naporafenib + trametinib to be studied in Stage 2 | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-254 and trametinib
Stage 1:To select the optimal dose of naporafenib + trametinib to be studied in Stage 2 | Study Day 1 up to Day 29
  Time to achieve maximum plasma concentration of ERAS-254 and trametinib
Stage 1:To select the optimal dose of naporafenib + trametinib to be studied in Stage 2 | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve
Stage 2: To compare PFS and OS for patients who are randomized to receive the combination of naporafenib + trametinib to that of patients who receive physician's choice of therapy (dacarbazine, temozolomide, or trametinib monotherapy) | Assessed up to 24 months from time of first dose
  * Progression free survival (PFS) based on assessment of radiographic imaging per RECIST v1.1
  * Survival status

SECONDARY OUTCOMES:
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs
Duration of Response (DOR) | Assessed up to 24 months from time of first dose]
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months from time of first dose]
  Based on assessment of radiographic imaging per RECIST version 1.1
Disease Control Rate (DCR) | Assessed up to 24 months from time of first dose]
  Based on assessment of radiographic imaging per RECIST version 1.1
Overall Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on the assessment of radiographic imaging per RECIST version 1.1
Plasma concentration (Cmax):Stage 1 only | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-254 and trametinib
Area under the curve (AUC):Stage 1 only | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve
Quality of Life: To assess disease and treatment-related QOL in patients with NRASm melanoma. | Assessed up to 24 months from time of first dose
  Using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire [QLQ]-C30 subscales and PRO CTCAE® symptom items specific to the potential cutaneous toxicities.

OTHER OUTCOMES:
Duration of Response (DOR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Overall Response Rate (ORR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)
Disease Control Rate (DCR) for CNS disease in participants | Assessed up to 24 months from time of first dose
  Based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Antal, Study Director — Clinical Development
Locations (59):
- United States (21):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - The Melanoma and Skin Care Institute, Englewood, Colorado
  - Mayo Clinic - Florida, Jacksonville, Florida
  - University of Miami Sylvester Cancer, Miami, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - SCRI Oncology Partners (formerly Tennessee Oncology), Nashville, Tennessee
  - Texas Oncology- Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Utah - Huntsman Cancer Institute (HCI), Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Tasman Health Care, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Institute, Melbourne, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Alfred Hospital, Melbourne
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McGill University Health Centre, Montreal, Quebec
- Czechia (3):
  - Masarykuv Onkologicky Ustav-MOU, Brno
  - Fakultni nemocnice Hradec Kralove, Nový Hradec Králové
  - Sanatorium Profesora Arenbergera, Prague
- France (9):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hospitalier Saint-Andre, Bordeaux
  - CHU Dijon Bourgogne - Hopital Francois Mitterand (Hopital du Bocage), Dijon
  - Centre Hospitalier du Mans, Le Mans
  - CHRU de Lille - HÃ´pital Claude Huriez, Lille
  - Centre Hospitalier Lyon-Sud, Lyon
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital de la Timone, Marseille
  - Hospital Ambroise Pairs, Paris
  - APHP - Hopital Saint Louis, Paris
  - CLCC Institute Gustave Roussy, Villejuif
- Italy (4):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario Sa, Milan
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Dermopatico dell Immacolata IDI-IRCCS, Roma
  - Azienda Sanitaria Universitaria del Friuli Centrale, Udine
- Netherlands (3):
  - Isala Ziekenhuis, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud University, Nijmegen
- Spain (6):
  - Hospital Universitari Vall d'Hebron - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (5):
  - Royal Preston Hospital, Preston, Lancashire
  - Sarah Cannon Research Institute - HCA Healthcare, City of London, London
  - Royal Devon and Exeter Hospital, Exeter
  - The Royal Marsden NHS Foundation Trust, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No